CLINICAL TRIAL: NCT03634553
Title: Evidence Based Training and Physical Activity With an E-health Program - a New Method for People With Chronic Obstructive Pulmonary Disease (COPD) to Become More Physically Active.
Brief Title: Evidence Based Training and Physical Activity With an E-health Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Alexandra Halvarsson, Principal Investigator, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-1738/2018
Record Dates: First submitted 2018-06-21; First posted 2018-08-16 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COPD; Physical Activity; Implementation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Training with e-health product The training program follows the recommendations for training from ACSMS and SoS who states the importance that exercise programs should include muscle strengthening, cardiovascular as wells as balance exercises. Therefore, the training program includes: Strengthening exercises for the upper and lower extremities (number: 5-8 pc. with progression in three levels), daily (5-7 times / week), 30 minutes walks and balance training.
  Interventions: Other: Training with e-health product
- Control (Active Comparator): usual care, i.e. participates in regular training regime at the physiotherapy department
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Training with e-health product — The training program follows the recommendations for training from ACSMS and SoS who states the importance that exercise programs should include muscle strengthening, cardiovascular as wells as balance exercises. Therefore, the training program includes: Strengthening exercises for the upper and lower extremities (number: 5-8 pc. with progression in three levels), daily (5-7 times / week), 30 minutes walks and balance training.
  Arms: Intervention
Other: Usual care — usual care, i.e. participates in regular training regime at the physiotherapy department
  Arms: Control

SUMMARY:
The main aim of the project in this application is two-fold. First we will explore and describe facilitators and barriers for being physically active and perform physical training for people with Chronic Obstructive Pulmonary Disease COPD (Step 1). Secondly, with user involvement, we will develop and evaluate a novel e-health program with a training module and an evidence-based educational component, the rEACH-COPD e-health program with the aim to increase the understanding and management of the disease and to facilitate every-day living with COPD (Step 2-3).

According to the guidelines of the Swedish National Board of Health and Welfare (SoS), physiotherapy led exercise is an important part of rehabilitation for people with COPD. The e-health training program will follow evidence-based guidelines, i.e. recommendations from SoS and the American College of Sport Medicine (ACSMS).

Offering individualized and evidence-based training will increase adherence to training. With regular physical activity and exercise there is a potential to improve health-related quality of life, physical capacity, activity and participation in every day life in people with COPD.

By an improved health, physical function and quality of life a decreased use of health care is expected. Thus, this program may, in the long term, contribute to reduced costs for the society.

DETAILED DESCRIPTION:
There is convincing evidence that physical activity and exercise have positive effects on quality of life and health in people with chronic disease and/or disabilities, but training programs do not reach all in need for it. Being able to offer individualized evidence-based training with modern technology (e-health) is an option, that may increase participation in health enhancing physical activity in people with chronic diseases.

The main aim of the project in this application is two-fold. First we will explore and describe facilitators and barriers for being physically active and perform physical training for people with Chronic Obstructive Pulmonary Disease COPD (Step 1). Secondly, with user involvement, we will develop and evaluate a novel e-health program with a training module and an evidence-based educational component, the rEACH-COPD e-health program with the aim to increase the understanding and management of the disease and to facilitate every-day living with COPD (Step 2-3).

Participants will be recruited from both Stockholm and Västerbotten county, university hospitals and primary care.

According to the guidelines of the Swedish National Board of Health and Welfare (SoS), physiotherapy led exercise is an important part of rehabilitation for people with COPD. The e-health training program will follow evidence-based guidelines, i.e. recommendations from SoS and the American College of Sport Medicine (ACSMS).

The e-health program will be developed and launched during 2019 and the participants will be included in the development to make the product feasible for the end users.

This project will contribute to improve health in people with COPD by using new technology.Offering individualized and evidence-based training will increase adherence to training. With regular physical activity and exercise there is a potential to improve health-related quality of life, physical capacity, activity and participation in every day life in people with COPD.

By an improved health, physical function and quality of life a decreased use of health care is expected. Thus, this program may, in the long term, contribute to reduced costs for the society.

Being able to offer training with an e-health program will give more people with COPD the opportunity to be physically active and thereby increase the chance for a better life with a good quality of life, less dependency in everyday life and add life to years and years to life. Physical activity and exercise offers a low-cost alternative with large health related effects which benefits both specific symptoms and general health in persons with COPD.

ELIGIBILITY:
Inclusion Criteria:

* participants must have a diagnosed COPD, be over 40 years and have no other medical barriers to participate in training at home with the e-health program.

Exclusion Criteria:

* medical barriers to participate in training at home with the e-health program.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test, CAT, to assess symtoms of COPD | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Questionnaire with 8 questions, graded 0-5. Total sum range from 0-40. High scores indicate high prevalence of symtoms.

SECONDARY OUTCOMES:
EuroQoL (EQ5D) assess health-related quality of life | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Questionnaire with 5 questions with 3 possible responses. The score are calculated with their own index list. The last question is a question with response option of a visual analog scale.
Leicester Cough Questionnaire LCQ-S assess health-related quality of life related to cough | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Questionnaire with 19 questions, graded 1-7. The score can be divided into three domains: physical, psychological and social. The domain sum is calculated by producing the average for each domain. These are then combined to give the total sum, which can vary from 3 to 21. Higher scores indicate better health related quality of life
mMRC (Medical Research Council Scale) assess symtoms of COPD | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  One scale ranging from 0-4, 4 indicate severe symtoms.
the Hospital anxiety and depression Scale, HAD, assess anxiety and depression | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Questionnaire with 14 questions, graded 0-4. Contains of two domains, anxiety and depression. Total score for each domain is calculated and higher scores indicates higher levels of anxiety or depression.
The SCI Exercise Self-Efficacy Scale assess Self-efficacy of their own ability to cope with physical activities | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Questionnaire with 10 questions, graded 1-4. Total score of 10-40, higher scores indicate higher ability
Frändin Grimby scale to assess Physical activity level | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  One scale ranging from 1-6, higher score indicate higher physical activity level
Accelerometer to assess physical activity level and pattern | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Accelerometer that assess different parameters related to physical activity pattern and level. Data collection during 5 days.
MiniBESTest asses balance performance | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Measurement consisting of 14 items, graded 0-2. The measurement consists of four domains and total score for each domain can be calculated and by sum up the domains a total score is given. Higher score indicate better balance performance
The Activities-specific Balance Confidence scale (ABC scale) assess balance confidence | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Questionnaire with 16 questions, graded 0-10. Total score is calculated by counting up all the 16 questions and thereafter divide by 16.
6-minute walk test to assess physical performance | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  walk test during 6 minutes. The total length is noted.
Sit to stand test to assess muscle strength in the lower leg. | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Number of rises from a chair are counted during 30 and 60 seconds.
10 meter walking test to assess walking speed. | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  The walking speed is calculated by taking time while the participant walk 10 meters during preferred and fast speed.
Hand grip test to assess hand grip strength | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Assess hand grip strength with a hand dynamometer.
Fall efficacy scale international (FES-I) to assess concerns about falling | Assess change from baseline to 10 weeks, 6 month and 12 month follow-up
  Questionnaire with 16 questions, graded 1-4. Total score of 16-64. Higher score indicate higher level of concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Halvarsson, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633